CLINICAL TRIAL: NCT02840383
Title: Participatory Trial of a Health Promoting School Approach to Positive Youth Development and Wellness Promotion
Brief Title: Trial of a Health Promoting School Approach to Positive Youth Development and Wellness Promotion
Acronym: TRUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); SoLaHmo (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1601S82061; 1U01MD010586-01 (NIH)
Record Dates: First submitted 2016-06-08; First posted 2016-07-21 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Adolescent School Connectedness; Adolescent Health; Community Based Participatory Research Methods
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Intervention (Active Comparator): Schools not receiving intervention until two years after implementation.
  Interventions: Other: Delayed Intervention
- Intervention (Experimental): Schools receiving intervention at the beginning of study.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Delayed Intervention — Schools not receiving intervention until two years after implementation.
  Arms: Delayed Intervention
Other: Intervention — intervention at the beginning of study.
  Arms: Intervention

SUMMARY:
Assess the effects of a school-based multi-component intervention on school connectedness, school engagement, and developmental assets through a group randomized, participatory trial.

DETAILED DESCRIPTION:
Health Promoting Schools intervention including pilot-tested teacher professional development, student-defined enhanced environment, and parent-defined enhanced community/family connection. The Coalition will finalize the intervention using a phased intervention map that integrates community perspectives with theoretical approaches to evidence based practices. The study aims will be accomplished through a group randomized trial in 10 urban schools with diverse populations representing approximately 1,900 students.

Aim 1: Assess the effects of a school-based multi-component intervention on school connectedness, school engagement, and developmental assets through a group randomized, participatory trial.

Hypothesis 1a: Students in the intervention schools will experience improved school connectedness, engagement and developmental assets compared to the control group.

Aim 2: Assess the effects of a school-based multi-component intervention on emotional well-being, tobacco and other substance use, and academic outcomes through a group randomized, participatory trial.

Hypothesis 2a: Students in the intervention schools will experience improved emotional well-being, course completion, attendance, and decreased disciplinary action and substance use compared to the control group.

Aim 3: Evaluate the relationships between participatory factors , school intervention implementation, and study outcomes.

Exploratory hypothesis 3a: Perceptions of quality of collaborative processes will be associated with degree of school intervention implementation and study outcomes.

Exploratory hypothesis 3b: School capacities and context will be associated with school intervention implementation and study outcomes.

Exploratory hypothesis 3c: School capacities and context will mediate the relationship between quality of collaborative processes and school intervention implementation.

ELIGIBILITY:
Inclusion Criteria:

* 9th grade students
* enrolled in the school at the time of randomization

Exclusion Criteria:

* Being unable to participate in the survey

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 811 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Baseline student school connectivity on a scale of 1-10 | 5 years
  Assess the effects of a school-based multi-component intervention on school connectedness, school engagement, and developmental assets through a group randomized, participatory trial.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Allen, MD, Principal Investigator — University of Minnesota, Department of Family Medicine
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided